CLINICAL TRIAL: NCT03636087
Title: Impact of an Enhanced Sterile Protocol on Root Canal Treatment Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: King's College London (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 242774
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Endodontic Disease; Root Canal Treatment; Root Canal Infection
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Root Canal Preparation; Root Canal Obturation

STUDY DESIGN:
Intervention Model Description: The study is single blind since the patient will not be aware of what technique is being used. The study cannot be double blind because the dentist will need to identify the protocol to follow. Randomization by blocks (block size 4) will be performed by a statistician at Kings College Dental Institute.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Access cavity preparation Working length determination Root canal instrumentation and chemo-mechanical preparation Root canal obturation Coronal restoration build up Cone Beam Computed Tomography scanning (CBCT) Radiographic imaging using periapical radiographs
  Interventions: Procedure: Access cavity preparation; Procedure: Working Length Determination; Procedure: Root canal instrumentation and chemo-mechanical preparation; Procedure: Root canal obturation; Procedure: Coronal restoration build up; Radiation: Cone Beam Computed Tomography scanning (CBCT); Radiation: Radiographic imaging using periapical radiographs
- Enhanced sterile protocol (Experimental): Access cavity preparation Working length determination Root canal instrumentation and chemo-mechanical preparation Root canal obturation Coronal restoration build up Changing gloves before obturation Disinfecting rubber dam The use of new instruments at time of obturation Cone Beam Computed Tomography scanning (CBCT) Radiographic imaging using periapical radiographs
  Interventions: Procedure: Access cavity preparation; Procedure: Working Length Determination; Procedure: Root canal instrumentation and chemo-mechanical preparation; Procedure: Root canal obturation; Procedure: Coronal restoration build up; Other: Changing gloves before obturation; Other: Disinfecting rubber dam; Other: The use of new instruments at time of obturation; Radiation: Cone Beam Computed Tomography scanning (CBCT); Radiation: Radiographic imaging using periapical radiographs

INTERVENTIONS:
Procedure: Access cavity preparation — High speed handpieces will be used with access burs to open the pulp chamber and get access to the root canal system (As a part of conventional root canal treatment established protocol)
Procedure: Working Length Determination — The length of the root canal will be measured using periodical radiographs and Electronic Apex Locators (As a part of conventional root canal treatment established protocol)
Procedure: Root canal instrumentation and chemo-mechanical preparation — Rotary files used to properly instrument and prepare canals length and size (As a part of conventional root canal treatment established protocol)
Procedure: Root canal obturation — Gutta Percha filling materials will be used to fill the root canal space with root canal sealer (As a part of conventional root canal treatment established protocol)
Procedure: Coronal restoration build up — A Build up material to seal the accessed tooth properly (As a part of conventional root canal treatment established protocol)
Other: Changing gloves before obturation — The treating dentist will change gloves before obturation
  Arms: Enhanced sterile protocol
Other: Disinfecting rubber dam — 2.25% Sodium Hypochlorite solution will be used to disinfect the rubber dam surface
  Arms: Enhanced sterile protocol
Other: The use of new instruments at time of obturation — A new instrument's kit will be use at the time of obturation
  Arms: Enhanced sterile protocol
Radiation: Cone Beam Computed Tomography scanning (CBCT) — CBCT will be taken before treatment and one year after completion
Radiation: Radiographic imaging using periapical radiographs — Periapical radiographs will be taken before, during and one year after the treatment completion (As a part of conventional root canal treatment established protocol)

SUMMARY:
The main goal of root canal treatment is the removal of existing microorganisms and the prevention of introducing new ones to the root canal system. This will require the application of strict aseptic measures. Microorganisms may also find their way into the root canal system through dental materials and instruments that are used during the treatment.

Some studies have suggested the necessity of decontamination of these materials and instruments prior to using. Also, the practice of changing gloves and disinfecting the tooth and rubber dam may help to reduce the possibility of introducing bacteria into the root canal space.

This study is aimed to evaluate the success rate of initial root canal treatment using an enhanced sterility protocol.

DETAILED DESCRIPTION:
Patients will be randomized to either group 1 or 2.Randomization by blocks will be performed by a statistician at Kings College Dental Institute. Group 1 will receive a conventional root canal therapy. While in group 2,clinician will follow sterile protocol. This will be carried out at KCL Dental Institute at Guy's Hospital as a part of the routine dental treatment at the endodontic postgraduate unit. Potential participants will be given a written information sheet and sufficient time to consider participation. Fully informed written consent will be obtained if they are interested in participation.

After providing consent, all participants will receive dental periapical (PA) radiograph and Cone Beam Computed Tomography (CBCT) scans which are part of standard care in root canal treatment. Then, a clinical assessment will be carried out for the tooth needing treatment which is routinely done before treatment.

Participants will then be randomly assigned to one of treatment groups. Treatment will be carried out by MclinDent postgraduate students (PG) supervised by their assigned clinical supervisor. It is a standard of care for PG students to undertake this type of treatment. During the treatment, clinical samples will be taken from tooth decay and from the root canal. These samples will undergo microbiological analysis by the research team.

After one year, all patients will be contacted for follow up appointment. Paired clinical and radiographic examination (PA and CBCT) will be carried out, matching the baseline measures. Healing will be evaluated radiographically and clinically. The tooth of interest will be examined for any pain or discomfort, the restoration will be evaluated, and the scans will be checked for radiographic healing. This follow up procedure is a standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients seeking root canal treatment over 18 years old.
2. Healthy patients.
3. Diagnosed with Irreversible pulpitis or pulpal necrosis on any molar tooth and accepting root canal treatment.

Exclusion Criteria:

1. Patients with clinical and radiographic diagnosis of previously treated root canal.
2. Anterior or premolar teeth.
3. Evidence of external or internal root resorption.
4. Pregnant women.
5. Patients younger than 18.
6. Patients unable to give consent.
7. Patients with compromised medical condition that affect the outcome of root canal therapy.
8. Non-restorable teeth.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-02 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical healing of root canal treated teeth | one year follow up after treatment completion
  Absence of symptoms reported by the patient.
Clinical healing of root canal treated teeth | one year follow up after treatment completion
  Absence of pain with Percussion test.
Clinical healing of root canal treated teeth | one year follow up after treatment completion
  Clinical examination to assess of the coronal filling.
Clinical healing of root canal treated teeth | one year follow up after treatment completion
  Clinical examination of the soft tissue integrity around treated tooth(Absence of bumps, lumps or swelling)

SECONDARY OUTCOMES:
Radiographic healing of root canal treated teeth with periapical radiographs | one year follow up after treatment completion
  Healing of the bony area around the root tip assessed by the absence or change in the size of radiolucincies (Darkness) in the x-rays.
Radiographic healing of root canal treated teeth with Cone Beam Computed Tompgraphy | one year follow up after treatment completion
  Healing of the bony area around the root tip assessed by the absence or change in the size of radiolucincies (Darkness) in the x-rays.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Mannocci, PhD, Principal Investigator — Professor of Endodontology and 1st Academic Supervisor
Locations (1):
- guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Consented patients will be allocated an a pseudo anonymized number. This number will be used for the sample collection and all study analysis.
  The Principal Investigator will maintain a document database of all patient's allocation numbers. Personal data, clinical notes and treatment records will be recorded in SALUD software as part of routine dental treatment at Guy's hospital. Only the chief investigator and supervisors will have access to the participants' allocation numbers and thus treatment records in SALUD during the study.